CLINICAL TRIAL: NCT06438393
Title: Screening Coronary Artery Disease Using artiFicial intelligencE in Non-contrast Computed Tomography
Acronym: SAFE-CT
Status: Not yet recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: University of Oxford (Other); University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: SAFE-CT
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Coronary Atheroscleroses
Keywords: Artificial intelligence; Radiomics; Deep learning; Coronary artery disease; Non-contrast computed tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples for proteomics analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stable chest pain and unknown CAD who underwent CTCA and CCS in the same scanning session: CAD: Presence of minimal coronary artery disease (i.e., coronary stenosis 0-25%) Normal coronary arteries: No visible coronary atherosclerosis
  Interventions: Diagnostic Test: CT coronary angiography and non-contrast CT

INTERVENTIONS:
Diagnostic Test: CT coronary angiography and non-contrast CT — A CTCA is an X-ray computed tomography of the coronary arteries that allows visualization of coronary plaques with high temporal and spatial resolution, however, it implies the use of iodine contrast and exposition to clinically significant ionizing radiation.
  Non-contrast ECG-gated CT ("calcium score" - CCS image). A non-contrast cardiac CT for CCS can be performed very quickly with significantly lower radiation (~6 times lower) than CTCA and without the need for contrast.
  Other Names: Non-contrast computed tomography

SUMMARY:
This project aims to improve direct patient care by reducing the risks of futile exposure to ionizing radiation and iodinated contrast in patients referred for coronary computed tomography angiography

DETAILED DESCRIPTION:
Since the last NICE guidelines update recommending computed tomography coronary angiography (CTCA) as the first line of investigation for patients with suspected coronary artery disease (CAD), there has been a high burden in the healthcare system and unnecessary exposition to radiation and iodine-containing contrast medium, especially in the youngest. Around 35% of patients who currently undergo CTCA have normal coronaries which means those patients were unnecessary exposed to radiation and contrast. A CTCA screening strategy to rule out CAD is needed to comply with the ALARA ("As Low As Reasonable Achievable") principles preventing radiation risks, reducing unnecessary scans and directing healthcare resources to those who will benefit from a CTCA.

We designed the SAFE-CT (Screening coronary Artery disease using artiFicial intelligencE in noncontrast Computed Tomography) study to develop a state-of-art artificial intelligence method to detect CAD as defined on CTCA using high-dimensional data (radiomics) extracted from the non-contrast cardiac computed tomography (CT). The model will be trained in 15,000 subjects scanned with paired non-contrast CT and CTCA and externally validated in an independent cohort of 1,000 subjects. In a preliminary analysis, non-contrast CT radiomics improved calcium score performance and discriminated CAD with an AUC of 0.91 (95% CI: 0.83-1.00). The algorithm will be converted into a user-friendly plugin to automatically decide whether the patient needs contrast. A real-world multicentre cohort study will be planned for software prospective validation and the creation of a large-scale proteomic biobank to support the translation of imaging biomarkers worldwide.

SAFE-CT can change the current CT scanning workflow by creating software that accurately rules out any CAD in >1/3 of patients referred for CTCA with low radiation and no contrast. This accurate machine learning model will be optimized to reach >90% sensitivity and negative predictive value and will bring several advantages for patients and the healthcare system:

* Prevention of radiation and contrast exposition.
* Increased CTCA scanning capacity for complex cases.
* Widespread use of CT for CAD exclusion in the emergency department and in outpatient clinics of centres with no CTCA.
* Improved screening tool for CAD in asymptomatic subjects.
* Up- and downstream cost reduction.

The SAFE-CT project proposes a safer, low-cost, and personalized CTCA scanning strategy that fosters scientific and technological innovation with the potential to bring improvement to patient care and clinical practice, and, thereby, societal, and economic impact.

ELIGIBILITY:
Inclusion Criteria:

- Patient with stable chest pain who underwent a CTCA

Exclusion Criteria:

* Missing non-contrast CT image (coronary calcium score image)
* Known coronary artery disease
* Prior myocardial infarction
* Prior PCI or CABG

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable chest pain patients with unknown CAD who underwent a CTCA with paired non-contrast CT
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Build a non-contrast CT radiomic signature of CAD | 3 years
Implement a machine learning model to discriminate patients with no CAD from patients with at least minimal disease (CAD-RADS=0 vs. CAD-RADS>0). | 3 years
Implement a machine learning model to detect coronary inflammation as defined using the Fat Attenuation Index (FAI ≥ -70.1 HU) in patients with no visible coronary plaque (CAD-RADS=0). | 3 years
Build a user-friendly plugin to facilitate users experience and distribution of our technology in clinical practice. | 3 years
Evaluate the real-world operationality and performance of the plugin in an international multicentre prospective cohort study. | 3 years
Create a national registry of cardiac CT | 3 years

SECONDARY OUTCOMES:
Setup a human blood biobank to identify the peripheral blood mononuclear cells (PBMCs) and plasma proteomics associated with CT data and clinical outcomes. | 3 years
Setup a public CT imaging repository | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided